CLINICAL TRIAL: NCT02199886
Title: A Phase I Single Dose-escalation Study of BIBH 1 in Patients With Non-small Cell Lung Cancer Scheduled for Surgical Resection
Brief Title: Dose-escalation Study of BIBH 1 in Patients With Non-small Cell Lung Cancer Scheduled for Surgical Resection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1152.3
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

ARMS (1):
- BIBH 1 (Experimental): dose escalation: 0.5, 2, 10 or 20mg/m**2, 7 days prior to surgery
  Interventions: Drug: BIBH 1

INTERVENTIONS:
Drug: BIBH 1 — labeled with eight to ten millicurie of 131I

SUMMARY:
Study to assess the toxicity, pharmacokinetics, biodistribution and imaging characteristics associated with increasing doses of 131I-BIBH 1, to compare the uptake of 131I-BIBH 1 in tumour to that of normal tissue in patients with non-small cell lung cancer and to measure human anti-human antibody (HAHA) concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary or secondary advanced non-small cell lung cancer
* Eligible for a lung biopsy or scheduled for surgery that would provide biopsy material
* Karnofsky performance status of ≥ 70
* Expected survival of ≥ 3 months
* Greater than or equal to 18 years of age
* Absolute granulocyte count ≥ 2.5 x 10**9/L
* Lymphocyte count > 0.7 x 10**9/L
* Platelet count ≥ 100 x 10**9/L
* Serum Creatinine ≤ 2.0 mg/dl (0.20 mmol/L)
* Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 3x upper limit of normal
* Total bilirubin < 2 mg/dl or 34µmol (SI unit equivalent)
* Ability to provide written informed consent

Exclusion Criteria:

* Active metastatic disease to the central nervous system, exhibited by new or enlarging lesions on CT or MRI scan or within 3 months of treatment (i.e., surgery or radiotherapy) for brain metastases
* Exposure to an investigational agent within four weeks of the BIBH 1 infusion
* Patients that are not fully recovered from surgery. Because of the potential binding of BIBH 1 to healing scars, patients with incomplete healing at an incision site, as evidenced by incomplete granulation, infection or localized edema are excluded
* Chemotherapy or immunotherapy within four weeks preceding entry (six weeks for nitrsoureas and/or mitomycin-C.)
* Previous administration of a murine, chimeric or humanised measurement and/or antibody fragment
* Serious illness: e.g., active infections requiring antibiotics, bleeding disorders or diseases considered by the investigator to have potential for interfering with obtaining accurate results from this study
* Women who are breast-feeding or pregnant
* Men and women of childbearing potential who are unwilling to utilize a medically acceptable method of contraception
* Previous participation in this study
* Patients who have autoimmune disease or hypertopic skin conditions that possibly over-express Fibroblast Activation Protein and may be targeted by the antibody. These diseases include active inflammatory arthritis, cirrhosis and keloids.
* Patients with unstable angina pectoris. Patients prescribed medication to control their angina pectoris must be on a fixed dose for at least 1 month prior to screening to be eligible for the trial.
* Patients who experienced a myocardial infarction within 3 months of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1998-07; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities as defined by Common toxicity criteria (CTC) | up to 30 days
Number of patients with abnormal biodistribution for 131I BIBH 1 | up to day 30
Tumor absorbed dose of 131I BIBH 1 | week 2

SECONDARY OUTCOMES:
Concentration of human anti-human antibodies (HAHA) | up to day 30